CLINICAL TRIAL: NCT05801341
Title: The Utility of "Lollipop" Oral Swabs in the Diagnosis of COVID-19 in an Inpatient Setting
Brief Title: Inpatient COVID-19 Lollipop Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lab evaluation of lollipop samples no longer available.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-0290; Protocol Version 4/4/2023 (Other: UW Madison); SMPH\PEDIATRICS\INFECT DIS (Other: UW Madison)
Record Dates: First submitted 2023-04-04; First posted 2023-04-06 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: COVID-19; Diagnostic Test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- COVID-19 Positive Participants (Experimental): Determined by NP PCR test
  Interventions: Device: Lollipop

INTERVENTIONS:
Device: Lollipop — An oral lollipop swab will be obtained by placing a flocked swab into the mouth and sucking on the swab for 20 seconds as one would suck on a lollipop
  Other Names: Lollipop collection swab

SUMMARY:
This study is being done to see if collecting saliva samples with a "lollipop" collection method works as well as nasopharyngeal samples for COVID-19 polymerase chain reaction (PCR) testing. 225 COVID-positive participants aged 4 years and above admitted to a hospital in the Madison, Wisconsin metropolitan area will be enrolled over a 6 month period.

DETAILED DESCRIPTION:
This is a prospective quantitative study evaluating the utility of a novel method of saliva collection for COVID-19 testing.

Primary Objective

* To determine the performance characteristics of oral lollipop swabs compared to Nasal Pharyngeal (NP) swabs for diagnosing COVID-19 via PCR molecular testing.

Secondary Objectives

* To identify clinical characteristics of patients when there are discordant results for NP and oral lollipop test results.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to provide verbal informed consent, if 18 years or older. If 4-17 years old, ability to understand and the willingness to provide verbal assent, plus have a parent or legal guardian present who can provide verbal informed consent.
* Willing to comply with all study procedures and be available for the duration of the study.
* Admitted to UW Health University Hospital or UW Health Kids American Family Children's Hospital.
* Individuals at least 4 years of age.
* Verified COVID-19 according to positive NP PCR test criteria.
* Enroll within 47 hours of the diagnostic NP swab; lollipop swab collected within 48 hours of the diagnostic NP swab.
* Either personally able or have a parent or legal guardian able to verbally answer questions in English about clinical symptoms, exposures, and other health and demographic information.

Exclusion Criteria:

* Unable to suck on a swab.
* Previous participation in this study.
* Require translation services for medical care.
* Not suitable for study participation due to other reasons at the discretion of the investigators or their designee.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Wald, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: COVID-19 positive participants were enrolled at UWHealth from April to May 2023.
Groups:
- COVID-19 Positive Participants: Participants were determined to be COVID-19 positive by NP PCR test for eligibility and subsequently tested for COVID-19 with Lollipop Swab PCR by placing a flocked swab into the mouth and sucking on the swab for 20 seconds as one would suck on a lollipop.
Period: Overall Study
Arm/Group | COVID-19 Positive Participants
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | COVID-19 Positive Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Tabulated Results From Nasopharyngeal (NP) vs Lollipop Swab-based PCR Covid-19 Tests
Description: Count of tests that detected COVID-19.
Time Frame: 1 study visit (data collected in 20 seconds)
Measure: Count of Units; unit: COVID-19 tests
Units Other Than Participants: COVID-19 tests
Groups:
- NP Swab Results: NP Swab PCR used to diagnose COVID-19 for eligibility.
- Lollipop Swab Results: Lollipop Swab sample collection device to test against gold-standard nasal swab PCR
Arm/Group | NP Swab Results | Lollipop Swab Results
Number analyzed (Participants) | 17 | 17
Number analyzed (COVID-19 tests) | 17 | 17
COVID-19 tests
  Covid-19 Detected | 17 | 4
  Covid-19 Not Detected | 0 | 13

2. Primary Outcome: Sensitivity: True Positive Rate
Description: NP vs. lollipop swab-based PCR COVID-19 tests. The True Positive Rate is the number of True Positive test results divided by the number of true positives and false negatives.
Time Frame: 1 study visit (data collected in 20 seconds)
Measure: Number; unit: percentage
Arm/Group | COVID-19 Positive Participants
Number analyzed (Participants) | 17
percentage | 23.5

3. Secondary Outcome: Number of Participants With Discordant Test Results
Description: All participants were confirmed COVID-19 positive by nasal-swab PCR test to be eligible for this study. Participants all took a COVID-19 test via lollipop-swab. Reported here are the number of participants who did not test positive for COVID-19 via the lollipop-swab device (discordant results).
Time Frame: 1 study visit (data collected in 20 seconds)
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Positive Participants
Number analyzed (Participants) | 17
Participants | 13

4. Secondary Outcome: Summary of COVID-19 Clinical Characteristics by Participant Count
Description: Count of participants who were: asymptomatic, symptomatic for less that 5 days, symptomatic for 5 days or greater, reported symptom days but ultimately determined to be asymptomatic by study team. Data collected via participant survey on the day of testing.
Time Frame: 1 study visit (data collected up to 15 minutes)
Population: 1 participant described symptoms that the study team determined were unrelated to COVID-19, and this participant is reported as asymptomatic here.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Positive Participants
Number analyzed (Participants) | 17
Participants
  Asymptomatic | 7
  Symptomatic for less than 5 days | 3
  Symptomatic for 5 days or greater | 7

5. Secondary Outcome: Summary of COVID-19 Clinical Characteristics by Discordant Results
Description: Of those with discordant results, how many were asymptomatic, symptomatic for less that 5 days, symptomatic for 5 days or greater, or reported symptom days but ultimately determined to be asymptomatic by study team. Data collected via participant survey on the day of testing.
Time Frame: 1 study visit (data collected in up to 10 minutes)
Population: Participants with discordant COVID-19 test results. 1 participant described symptoms that the study team determined were unrelated to COVID-19, and this participant is reported as asymptomatic here.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Positive Participants
Number analyzed (Participants) | 13
Participants
  Asymptomatic | 7
  Symptomatic for less than 5 days | 2
  Symptomatic for 5 days or greater | 4

ADVERSE EVENTS:
Time Frame: AEs were collected after the signing of consent until study procedures were completed (survey and sample collection, up to 15 minutes).
Arm/Group | COVID-19 Positive Participants
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
Statistical Analyses were not completed as planned because of premature termination. Participant population were patients with a positive PCR screening test at the time of admission to the hospital regardless of their history of acute respiratory symptoms. Study not powered per protocol for meaningful results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT05801341/Prot_SAP_000.pdf